CLINICAL TRIAL: NCT02353429
Title: Toremifene in Desmoid Tumor: Prospective Clinical Trial and Identification of Potential Molecular Targets
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 112/11
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Desmoid Type-fibromatosis
MeSH Terms: conditions — Desmoid Tumors | interventions — Toremifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Toremifene treatment (Experimental): Patients will receive 60 mg daily of Toremifene and the dose will be escalated to 180 mg daily in case of progression
  Interventions: Drug: Toremifene

INTERVENTIONS:
Drug: Toremifene — Patients will receive 60 mg daily and then 180 daily in case of progression

SUMMARY:
This is a prospective study evaluating the activity and the safety of toremifene in patients with primary or recurrent sporadic DTs.

Patients will be enrolled after the histological confirmation of DTs on biopsy Patients will start at 60 mg daily and dose-escalate to 180 mg upon progression. Disease assessment will be performed by contrast-enhanced MRI or CT scan, pain evaluation by a visual analog scale (VAS) every 3 months for the first and second year, twice yearly thereafter. Response will be evaluated either by RECIST and/or symptomatic relief.

DETAILED DESCRIPTION:
This is a prospective study evaluating the activity and the safety of toremifene in patients with primary or recurrent sporadic DTs.

Patients will be enrolled after the histological confirmation of DTs on biopsy performed at the investigators institution or after the pathological review of tissue specimen obtained via needle biopsy or surgical excision (in case of recurrence) performed elsewhere. A new biopsy will be performed if the amount of tissue will not be sufficient for immunohistochemical analysis. Patients will start at 60 mg daily and dose-escalate to 180 mg upon progression. Disease assessment will be performed by contrast-enhanced MRI or CT scan, pain evaluation by a visual analog scale (VAS) every 3 months for the first and second year, twice yearly thereafter. Response will be evaluated either by RECIST and/or symptomatic relief.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years) with primary or locally recurrent, sporadic or FAP associated, desmoid fibromatosis
* Histologically documented diagnosis of DF
* At least one measurable site of disease at CT or MRI scans, which has not been previously embolised or irradiated
* Progressive disease demonstrated at contrast-enhanced MRI or CT scan by Response Evaluation Criteria in Solid Tumors (RECIST)
* Radiologic or clinical evidence of PD in the previous 6 months. Radiologic PD will be defined according to RECIST
* ECOG Performance status: 0-2
* Prior hormonal therapy, chemotherapy, or molecular targeted therapies are allowed
* Adequate end organ function, defined as the following: total bilirubin < 1.5 x ULN, SGOT and SGPT < 2.5 x UNL (or < 5 x ULN if hepatic metastases are present), creatinine < 1.5 x ULN, ANC > 1.5 x 109/L, platelets > 100 x 109/L
* Female patients of child-bearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug
* Life expectancy of at least 6 months
* Written, voluntary, informed consent.

Exclusion Criteria:

* Previous history of deep vein thrombosis
* Evidence of prolonged QTc >480 msec (using Bazetts correction, for which the formula is: QTc = QT/√RR) or history of familial long QT syndrome
* Previous arrhythmia
* Clinically significant bradycardia
* Endometrial hyperplasia
* Hepatic insufficiency
* Other concurrent hormonal therapy, including hormonal contraceptives
* Patient has received any other investigational agents within 28 days of first day of study drug dosing. - Female patients who are pregnant or breast-feeding
* Patient has a severe and/or uncontrolled medical disease
* Patient has a known diagnosis of human immunodeficiency virus (HIV) infection
* Patient received chemotherapy within 4 weeks prior to study entry
* Patient had a major surgery within 2 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Time to progression | 2 years
  This study evaluates clinical benefit by comparing sequentially measured paired failure times within each treated patient, namely time to progression after the 60 mg toremifene dose (TTP1) versus the (possibly censored) time to progression after the 180 mg toremifene dose (TTP2)

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Colombo, MD, Principal Investigator — Fondazione IRCCS Istituto Tumori Milano
Locations (1):
- Fondazione IRCCS Istituto Tumori Milano, Milan, Italy

REFERENCES:
- [Derived] Fiore M, Colombo C, Radaelli S, Callegaro D, Palassini E, Barisella M, Morosi C, Baldi GG, Stacchiotti S, Casali PG, Gronchi A. Hormonal manipulation with toremifene in sporadic desmoid-type fibromatosis. Eur J Cancer. 2015 Dec;51(18):2800-7. doi: 10.1016/j.ejca.2015.08.026. Epub 2015 Nov 18. PMID 26602014